CLINICAL TRIAL: NCT06316609
Title: Prenatal Exposure to Emerging Contaminants and Offspring's Atopic Dermatitis (PECCAD)
Brief Title: Prenatal Exposure to Emerging Contaminants and Children's Atopic Dermatitis
Acronym: PECCAD
Status: Active, not recruiting | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Collaborators: Minhang Maternal and Children Health Care Hospital (Other); School of Public Health，Fudan University (Unknown)
Responsible Party: Sponsor
Other Study IDs: AD2016-2027
Record Dates: First submitted 2024-02-27; First posted 2024-03-18 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Atopic Dermatitis
Keywords: Skin barrier; Microplastics; Organophosphate Flame Retardants, OPFRs; Perfluoroalkyl and Polyfluoroalkyl Substances, PFASs; Contaminants of Emerging Concern, CECs; Emerging Contaminants, ECs; Atopic Dermatitis; Maternal; Cohort; Birth
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — All serum, whole blood, and DNA samples are stored in a -80°C freezer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- participants from birth cohort with AD: The association between maternal whole blood and serum levels of Emerging Contaminants (ECs) including Per- and Polyfluoroalkyl Substances (PFASs), Organophosphate Flame Retardants (OPFRs), and Microplastics during pregnancy and the incidence of atopic dermatitis in their offspring.
  Interventions: Other: Gestational Exposure to Emerging Contaminants (ECs)
- participants from birth cohort without AD: The association between maternal whole blood and serum levels of Emerging Contaminants (ECs) including Per- and Polyfluoroalkyl Substances (PFASs), Organophosphate Flame Retardants (OPFRs), and Microplastics during pregnancy and the reduced incidence of atopic dermatitis in their offspring.
  Interventions: Other: Gestational Exposure to Emerging Contaminants (ECs)

INTERVENTIONS:
Other: Gestational Exposure to Emerging Contaminants (ECs) — Levels of Emerging Contaminants (ECs), such as Per- and Polyfluoroalkyl Substances (PFASs), Organophosphate Flame Retardants (OPFRs), and Microplastics, are assessed in maternal blood and umbilical cord blood during gestation.
  Other Names: Gestational Exposure to Contaminants of Emerging Concern (CECs); Gestational Exposure to Contaminants of Emerging pollutants

SUMMARY:
This prospective cohort study aims to investigate the association between prenatal blood levels of Emerging Contaminants and the five-year incidence of atopic dermatitis (AD) in offspring.

DETAILED DESCRIPTION:
This prospective birth cohort study, conducted within the Shanghai prenatal population, involves the collection of maternal blood samples during gestation to directly measure the biological exposure levels of Emerging Contaminants, including Per- and Polyfluoroalkyl Substances (PFAS), Organophosphate Flame Retardants (OPFRs), and Microplastics. Serum and whole blood levels of these contaminants are evaluated during pregnancy at 12-14, 22-26, and 31-34 gestational weeks. Subsequently, the study assesses skin barrier function in infants at 24-48 hours, 42 days, and 6 months of age. During a five-year period, the occurrence of atopic dermatitis (AD) in offspring is assessed. The objectives of this cohort study are twofold: (1) to elucidate the relationship between maternal exposure to Emerging Contaminants and the development of AD in offspring, and (2) to evaluate the impact of such exposure on the skin barrier function of infants. This research aims to provide substantial evidence for the prevention of AD, offering a unique and meaningful approach to mitigating the incidence of AD.

ELIGIBILITY:
Inclusion Criteria:

* Mother plans to proceed prenatal care and delivery in Minhang Maternal and Children Health Care Hospital
* 12-14 weeks of singleton pregnancy, non-stillborn or miscarrying, offspring without familial hereditary skin diseases
* Offspring plans to stay in Shanghai until 5 years and proceed follow-up at the Dermatology Department of Children's Hospital affiliated with Fudan University
* signed informed consent.

Exclusion Criteria:

* Multiple pregnancies
* perinatal death
* a fetus with congenital skin or appendages disorders

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The research subjects come from the established MKNFOAD birth cohort (NCT 02889081), with on-site inclusion at the early pregnancy outpatient clinic of Minhang Maternal and Child Health Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 456 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
atopic dermatitis: Infant atopic dermatitis incidence | at 1 year old
  Disease diagnosis according to the criteria of Williams. Skin status was examined via onsite interview by pediatric dermatologists. Parents consulted or visited a dermatologist once their baby developed any skin symptoms.

SECONDARY OUTCOMES:
atopic dermatitis | incidence of AD during 6 months after birth
  Disease diagnosis according to the criteria of Williams. Skin status was examined via onsite interview by pediatric dermatologists. Parents consulted or visited a dermatologist once their baby developed any skin symptoms.
atopic dermatitis | incidence of AD at the age of two.
  Disease diagnosis according to the criteria of Williams. Skin status was examined via onsite interview by pediatric dermatologists. Parents consulted or visited a dermatologist once their baby developed any skin symptoms.
atopic dermatitis | incidence of AD at the age of five.
  Disease diagnosis according to the criteria of Williams. Skin status was examined via onsite interview by pediatric dermatologists. Parents consulted or visited a dermatologist once their baby developed any skin symptoms.
prenatal exposure to Perfluoroalkyl and Polyfluoroalkyl Substances (PFASs) at early pregnancy | 12-14 gestational weeks
  Maternal whole blood levels of Perfluoroalkyl and Polyfluoroalkyl Substances (PFASs) comprising 15 variants: PFPeA, PFHxA, PFHpA, PFOA, PFNA, PFDA, PFUnDA, PFDoDA, PFTrDA, PFHpDA, PFBS, PFPeS, PFHxS, PFOS, and PFDS
prenatal exposure to Perfluoroalkyl and Polyfluoroalkyl Substances (PFASs) at mid pregnancy | 22-26 gestational weeks
  Maternal whole blood levels of Perfluoroalkyl and Polyfluoroalkyl Substances (PFASs) comprising 15 variants: PFPeA, PFHxA, PFHpA, PFOA, PFNA, PFDA, PFUnDA, PFDoDA, PFTrDA, PFHpDA, PFBS, PFPeS, PFHxS, PFOS, and PFDS
prenatal exposure to Perfluoroalkyl and Polyfluoroalkyl Substances (PFASs) at late pregnancy | 34-36 gestational weeks
  Maternal whole blood levels of Perfluoroalkyl and Polyfluoroalkyl Substances (PFASs) comprising 15 variants: PFPeA, PFHxA, PFHpA, PFOA, PFNA, PFDA, PFUnDA, PFDoDA, PFTrDA, PFHpDA, PFBS, PFPeS, PFHxS, PFOS, and PFDS
prenatal exposure to Perfluoroalkyl and Polyfluoroalkyl Substances (PFASs) at first trimester | 12-14 gestational weeks
  Maternal serum levels of Perfluoroalkyl and Polyfluoroalkyl Substances (PFASs) comprising 15 variants: PFPeA, PFHxA, PFHpA, PFOA, PFNA, PFDA, PFUnDA, PFDoDA, PFTrDA, PFHpDA, PFBS, PFPeS, PFHxS, PFOS, and PFDS
prenatal exposure to Perfluoroalkyl and Polyfluoroalkyl Substances (PFASs) at second trimester | 22-26 gestational weeks
  Maternal serum levels of Perfluoroalkyl and Polyfluoroalkyl Substances (PFASs) comprising 15 variants: PFPeA, PFHxA, PFHpA, PFOA, PFNA, PFDA, PFUnDA, PFDoDA, PFTrDA, PFHpDA, PFBS, PFPeS, PFHxS, PFOS, and PFDS
prenatal exposure to Perfluoroalkyl and Polyfluoroalkyl Substances (PFASs) at third trimester | 34-36 gestational weeks
  Maternal serum levels of Perfluoroalkyl and Polyfluoroalkyl Substances (PFASs) comprising 15 variants: PFPeA, PFHxA, PFHpA, PFOA, PFNA, PFDA, PFUnDA, PFDoDA, PFTrDA, PFHpDA, PFBS, PFPeS, PFHxS, PFOS, and PFDS
Perfluoroalkyl and Polyfluoroalkyl Substances (PFASs) in Umbilical cord whole blood | at delivery
  Umbilical cord whole blood levels of PFDoDA, PFTrDA, PFHpDA, PFBS, PFPeS, PFHxS, PFOS, and PFDS
Umbilical cord serum Perfluoroalkyl and Polyfluoroalkyl Substances (PFASs) | at delivery.
  Umbilical cord serum levels of PFDoDA, PFTrDA, PFHpDA, PFBS, PFPeS, PFHxS, PFOS, and PFDS
prenatal exposure to Organophosphate Flame Retardants (OPFRs) at early pregnancy | 12-14 gestational weeks
  Maternal whole blood levels of Organophosphate Flame Retardants (OPFRs) comprising 9 variants: TEP、TBP、TBEP/TBOEP、TPrP、TCEP、TCPP/TCIPP、TDCPP/TDCIPP、TDBP/TDBPP、TPhP/TPHP
prenatal exposure to Organophosphate Flame Retardants (OPFRs) at mid pregnancy | 22-26 gestational weeks
  Maternal whole blood levels of Organophosphate Flame Retardants (OPFRs) comprising 9 variants: TEP、TBP、TBEP/TBOEP、TPrP、TCEP、TCPP/TCIPP、TDCPP/TDCIPP、TDBP/TDBPP、TPhP/TPHP
prenatal exposure to Organophosphate Flame Retardants (OPFRs) at late pregnancy | 34-36 gestational weeks
  Maternal whole blood levels of Organophosphate Flame Retardants (OPFRs) comprising 9 variants: TEP、TBP、TBEP/TBOEP、TPrP、TCEP、TCPP/TCIPP、TDCPP/TDCIPP、TDBP/TDBPP、TPhP/TPHP
prenatal exposure to Organophosphate Flame Retardants (OPFRs) at first trimester | 12-14 gestational weeks
  Maternal serum levels of Organophosphate Flame Retardants (OPFRs) comprising 9 variants: TEP、TBP、TBEP/TBOEP、TPrP、TCEP、TCPP/TCIPP、TDCPP/TDCIPP、TDBP/TDBPP、TPhP/TPHP
prenatal exposure to Organophosphate Flame Retardants (OPFRs) at second trimester | 22-26 gestational weeks
  Maternal serum levels of Organophosphate Flame Retardants (OPFRs) comprising 9 variants: TEP、TBP、TBEP/TBOEP、TPrP、TCEP、TCPP/TCIPP、TDCPP/TDCIPP、TDBP/TDBPP、TPhP/TPHP
prenatal exposure to Organophosphate Flame Retardants (OPFRs) at third trimester | 34-36 gestational weeks
  Maternal serum levels of Organophosphate Flame Retardants (OPFRs) comprising 9 variants: TEP、TBP、TBEP/TBOEP、TPrP、TCEP、TCPP/TCIPP、TDCPP/TDCIPP、TDBP/TDBPP、TPhP/TPHP
Organophosphate Flame Retardants (OPFRs) in Umbilical cord whole blood | at delivery
  Umbilical cord whole blood levels of PFDoDA, PFTrDA, PFHpDA, PFBS, PFPeS, PFHxS, PFOS, and PFDS
Umbilical cord serum Organophosphate Flame Retardants (OPFRs) | at delivery
  Umbilical cord serum levels of PFDoDA, PFTrDA, PFHpDA, PFBS, PFPeS, PFHxS, PFOS, and PFDS
Infant skin barrier function (Transepidermal Water Loss, TEWL） | infant 24-48 hours
  TEWL will be evaluated by the device of Multi Probe Adapter 4.
Infant skin barrier function (Transepidermal Water Loss, TEWL） | infant 42 days old
  TEWL will be evaluated by the device of Multi Probe Adapter 4.
Infant skin barrier function (Transepidermal Water Loss, TEWL） | infant 6 months old
  TEWL will be evaluated by the device of Multi Probe Adapter 4.
Infant skin barrier function (Stratum corneum hydration, SCH) | infant 24-48 hours
  SCH will be evaluated by the device of Multi Probe Adapter 4.
Infant skin barrier function (Stratum corneum hydration, SCH) | infant 42 days old
  SCH will be evaluated by the device of Multi Probe Adapter 4.
Infant skin barrier function (Stratum corneum hydration, SCH) | infant 6 months old
  SCH will be evaluated by the device of Multi Probe Adapter 4.
Infant skin barrier function (sebum content) | infant 24-48 hours
  Sebum content will be evaluated by the device of Multi Probe Adapter 4.
Infant skin barrier function (sebum content) | infant 42 days old
  Sebum content will be evaluated by the device of Multi Probe Adapter 4.
Infant skin barrier function (sebum content) | infant 6 months old
  Sebum content will be evaluated by the device of Multi Probe Adapter 4.
Infant skin barrier function (skin surface pH) | infant 24-48 hours
  Skin pH will be evaluated by the device of Multi Probe Adapter 4.
Infant skin barrier function (skin surface pH) | infant 42 days old
  Skin pH will be evaluated by the device of Multi Probe Adapter 4.
Infant skin barrier function (skin surface pH) | infant 6 months old
  Skin pH will be evaluated by the device of Multi Probe Adapter 4.
prenatal exposure to Microplastics at early pregnancy | 12-14 gestational weeks
  Maternal whole blood levels of Microplastics
prenatal exposure to Microplastics at mid pregnancy | 22-26 gestational weeks
  Maternal whole blood levels of Microplastics
prenatal exposure to Microplastics at late pregnancy | 34-36 gestational weeks
  Maternal whole blood levels of Microplastics
prenatal exposure to Microplastics at first trimester | 12-14 gestational weeks
  Maternal serum levels of Microplastics
prenatal exposure to Microplastics at second trimester | 22-26 gestational weeks
  Maternal serum levels of Microplastics
prenatal exposure to Microplastics at third trimester | 34-36 gestational weeks
  Maternal serum levels of Microplastics
Microplastics in Umbilical cord whole blood | at delivery.
  Umbilical cord whole blood levels of Microplastics
Umbilical cord serum Microplastics | at delivery.
  Umbilical cord serum levels of Microplastics
Allergic rhinitis | incidence of allergic rhinitis at the age of five.
  An inquiry into the patient's medical history and electronic medical record
Asthma | incidence of asthma at the age of five.
  An inquiry into the patient's medical history and electronic medical record
Infantile hemangioma | incidence of Infantile hemangioma at 1 year old
  Diagnosed by dermatologists

CONTACTS AND LOCATIONS:
Overall Officials: Ying Ye, MD,PhD, Principal Investigator — Children's Hospital of Fudan University Shanghai, China, 201102
Locations (1):
- Children Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] Lowe AJ, Dharmage SC, Abramson MJ, Vijayasarathy S, Erbas B, Mueller JF, Lodge CJ. Cord-serum per- and poly-fluoroalkyl substances and atopy and eczema at 12-months. Allergy. 2019 Apr;74(4):812-815. doi: 10.1111/all.13669. Epub 2018 Dec 4. No abstract available. PMID 30428139
- [Background] Chen Q, Huang R, Hua L, Guo Y, Huang L, Zhao Y, Wang X, Zhang J. Prenatal exposure to perfluoroalkyl and polyfluoroalkyl substances and childhood atopic dermatitis: a prospective birth cohort study. Environ Health. 2018 Jan 17;17(1):8. doi: 10.1186/s12940-018-0352-7. PMID 29343261
- [Background] Okada E, Sasaki S, Kashino I, Matsuura H, Miyashita C, Kobayashi S, Itoh K, Ikeno T, Tamakoshi A, Kishi R. Prenatal exposure to perfluoroalkyl acids and allergic diseases in early childhood. Environ Int. 2014 Apr;65:127-34. doi: 10.1016/j.envint.2014.01.007. Epub 2014 Jan 29. PMID 24486970